CLINICAL TRIAL: NCT04058327
Title: A Study on Early Diagnosis and Treatments of Minimal Hepatic Encephalopathy(MHE) in Patients With Liver Diseases
Brief Title: A Study of MHE in Patients With Liver Diseases
Status: Completed | Type: Observational
Sponsor: Qin Ning (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, Director of Department of Infectious Diseases, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: MHE study
Record Dates: First submitted 2019-08-11; First posted 2019-08-15 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Hepatic Encephalopathy; Minimal Hepatic Encephalopathy; Overt Hepatic Encephalopathy
Keywords: neurophysiologica tests; diagnosis; minimal hepatic encephalopathy; overt hepatic encephalopathy; liver cirrhosis; acute on chronic liver failure; blood biomarkers
MeSH Terms: conditions — Hepatic Encephalopathy; Disease; Liver Cirrhosis; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma will be restored in central lab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MHE group: Patients whose MHE test are positive
  Interventions: Diagnostic Test: neurophysiological tests, blood biomarkers.
- no HE group: Patients whose MHE test are negative
  Interventions: Diagnostic Test: neurophysiological tests, blood biomarkers.

INTERVENTIONS:
Diagnostic Test: neurophysiological tests, blood biomarkers. — Let the patients do neuropsychological tests and detect blood biomarkers.

SUMMARY:
The study analyzes the diagnostic efficacy of neurophysiological tests and blood biomarkers on MHE, predicts risk factors on the development of OHE and investigate the mortality of MHE in patients with cirrhosis and acute on chronic liver failure.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a common complication and one of the most serious manifestations of cirrhosis and acute on chronic liver failure, not only increasing the risks of death, but also seriously affecting the lives of the patients and their caregivers. Minimal hepatic encephalopathy (MHE), the earliest stage of HE, despite its undiscernible clinical evidence, it is related with abnormalities of patients' daily cognition, emotion, muscular strength, driving ability, quality of life and socioeconomic status At present. However, MHE is not easy to diagnose in daily clinical work because of time-consuming psychometric tests, especially the inconvenience of application in weak inpatients. This study aims to analyze the diagnostic efficacy of neurophysiological tests and blood biomarkers on MHE, predict risk factors on the development of OHE and investigate the mortality of MHE in patients with cirrhosis and acute on chronic liver failure.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* cirrhosis
* acute on chronic liver failure

Exclusion Criteria:

(1) status of OHE; (2) accompanying nervous system diseases, such as dementia or stroke; (3) a history of recent head trauma or surgery, and (4) organic lesions in the brain, such as haemorrhages or infarction; (5) inability to finish the psychometric hepatic encephalopathy score (PHES), such as unable to observe patterns or words clearly on paper, and (6) a recent transjugular intrahepatic portosystemic shunt (TIPS) or abdominal imaging demonstrated portosystemic shunts, and (7) high alcohol consumption (> 30 g/day in men or 20 g/day in women) or psychoactive medication consumption in the past four weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis, acute on chronic liver failure
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
progression of 2-4 HE | 30 days
  Incidence of HE progression (2/3/4 HE)
mortality in short, median and long term | 30 and 90 days, 1, 2, 3 years
  mortality in 30 days, 90 days, 1 year, 2 years, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, MD., PhD., Study Chair — Department of Infectious Disease, Tongji Hospital, Tongji Medical College, HUST
Locations (1):
- Department of Infectious Disease, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China